CLINICAL TRIAL: NCT02730728
Title: A Randomized Study of Single Shot vs 24hr vs 48hr Continuous Adductor Canal Block for Postoperative Analgesia After Total Knee Arthroplasty
Brief Title: Single Shot vs 24hr vs 48hr Continuous Adductor Canal Block After TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 823219
Record Dates: First submitted 2016-03-23; First posted 2016-04-06 (Estimated); Results first posted 2018-06-18 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-05

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis; Post Operative Pain Control
Keywords: adductor canal block; tinetti score; time to up and go test; Ambulation distance; pain score; quality of recovery score
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single shot adductor canal block (Active Comparator): adductor canal block group will receive single shot adductor canal block with 20ml bolus of 0.5% ropivicaine for analgesia after TKA
  Interventions: Drug: 20ml bolus of 0.5% ropivicaine
- 24 hour continuous adductor canal block (Active Comparator): adductor canal block group will receive 24 hour continuous adductor canal block (0.2% Ropivicaine at 8 milliliter/hour) with initial 5ml bolus of 0.5% Ropivicaine for analgesia after TKA
  Interventions: Drug: 0.2% Ropivicaine at 8 milliliter/hour; Drug: 5ml bolus of 0.5% ropivicaine
- 48 hour continuous adductor canal block (Active Comparator): adductor canal block group will receive 48 hour continuous adductor canal block (0.2% Ropivicaine at 8 milliliter/hour) with initial 5ml bolus of 0.5% Ropivicaine for analgesia after TKA
  Interventions: Drug: 0.2% Ropivicaine at 8 milliliter/hour; Drug: 5ml bolus of 0.5% ropivicaine

INTERVENTIONS:
Drug: 20ml bolus of 0.5% ropivicaine — Local anesthetic
  Arms: Single shot adductor canal block
Drug: 0.2% Ropivicaine at 8 milliliter/hour — Local anesthetic
  Arms: 24 hour continuous adductor canal block; 48 hour continuous adductor canal block
Drug: 5ml bolus of 0.5% ropivicaine — Local anesthetic
  Arms: 24 hour continuous adductor canal block; 48 hour continuous adductor canal block

SUMMARY:
The purpose of this study is to compare a single shot block, 24 hours, and 48 hour continuous catheter nerve block done via the adductor canal method in adult patients who have under gone total knee arthroplasty. Visual analogue scores, opioid consumption, time to up and go, ambulation, manual muscle tests, and Tinetti scores up to 72 hours post operatively will be used for comparison.

DETAILED DESCRIPTION:
If the patient is willing to participate and signs the consent, he/she will be randomized to one of the three treatment groups:

1. Single shot block
2. 24 hour catheter
3. 48 hour catheter

The choice of anesthetic technique will be at the discretion of the anesthesiologist. In our institution we usually advocate for spinal anesthesia for total knee arthroplasty. All patients will receive their multimodal perioperative pain protocol (MP3) medication as per protocol in the patient receiving area (400 mg of gabapentin, 200 mg of Celecoxib, and 1gm of acetaminophen).

Patients will be monitored during block performance with standard ASA monitors. All patients will be receiving 2 L of oxygen via a nasal cannula. Sedatives will be titrated to effect. Midazolam 1-2 mg, and fentanyl 50-100 mcg will be used for sedation.

Block time out will be preformed according to standard operating procedure. All blocks will be done under ultrasound guidance. Sonosite S nerve machine will be used with a high frequency linear (HFL) US probe with 6-13 MHZ frequency. Both single shot and continuous adductor canal block will be performed according to the standard operating practices in our department 4. Ultrasound survey at the medial part of the thigh will take place, halfway between the superior anterior iliac spine and the patella. In a short axis view, the femoral artery will be identified underneath the sartorius muscle, with the vein just inferior and the saphenous nerve just lateral to the artery. The needle will be introduced in-plane and 2 to 3 mL of local anesthesia bolus will be used to verify correct placement of the needle in the vicinity of the saphenous nerve in the adductor canal.

For single shot blocks: A bolus of total volume of 20 ml of ropivicaine 0.5% will be injected through the needle.

For the continuous block: The catheter will be introduced and advanced 2-3 cm beyond the tip of the needle under ultrasound visualization. The needle was withdrawn over the catheter. Injection of a bolus of 5 ml of ropivacaine 0.5% will take place through the catheter while observing the spread of local anesthetic under ultrasound. The catheter hub will be affixed to the upper lateral thigh with sterile occlusive dressings and an anchoring device.

Block success will be defined as a change in cutaneous sensation to touch with an alcohol pad in the saphenous nerve distribution over the medial leg within 30min after injection. Subjects with successful catheter placement per protocol and nerve block onset were retained in the study. Subjects with a failed catheter insertion or misplaced catheter indicated by a lack of sensory changes had their catheter replaced or were withdrawn from the study.

At the conclusion of surgery, the catheters will be connected to a pump that will infuse local anesthetic. Ropivicaine 0.2% at 8 ml/hour. In the postoperative anesthesia care unit, intermittent boluses of hydromorphone will be used as needed. Postoperative analgesia will follow the MP3 protocol. Drugs that are used for the multimodal analgesia protocol include acetaminophen (1 gm every 8 hours for 72 hours), celecoxib (200 mg every 8 hours for 72 hours), Gabapentin (300 mg every 8 hours for one week if the patient is opioid naïve and for two weeks if patients are opioid tolerant), and oxycodone (5-10-15 mg oral as needed every 4 hours for pain based on patient reported pain score).

All patients will receive prophylaxis for postoperative nausea and vomiting (PONV) during surgery. The protocol for prophylaxis against PONV include administration of 4 mg of dexamethasone after induction of anesthesia and 4 mg of ondansetron 20 minutes before recovery from anesthesia. Dexamethasone is withheld if the patient has poorly controlled diabetes mellitus (DM). Uncontrolled DM will be defined as random blood glucose above 250 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary total knee arthroplasty
* American Society of Anesthesiologists (ASA) physical status I -III
* mentally competent and able to give consent for enrollment in the study

Exclusion Criteria:

* Patient younger than 18 years old
* Allergy to local anesthetics, systemic opioids (fentanyl, morphine, hydromorphone, and any of the drugs included in the multimodal perioperative pain protocol (MP3)
* Revision surgery
* Impaired kidney functions and patient with coagulopathy
* Chronic pain syndromes; Patients will be defined to have chronic pain if they are using regular daily doses of systemic narcotics for the past 3 months prior to the surgery
* BMI of 40 or more
* Pregnancy (positive urine pregnancy test result in Preop area on morning of surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M Elkassabany, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Shot Adductor Canal Block | 24 Hour Continuous Adductor Canal Block | 48 Hour Continuous Adductor Canal Block
Started | 53 | 53 | 53
Completed | 53 | 51 | 52
Not Completed | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Shot Adductor Canal Block | 24 Hour Continuous Adductor Canal Block | 48 Hour Continuous Adductor Canal Block | Total
Number analyzed (Participants) | 53 | 51 | 52 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.6) | 66.5 (8.5) | 62.2 (8.7) | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 18 | 56
  Male | 37 | 29 | 34 | 100

OUTCOME MEASURES:

1. Primary Outcome: Patients With Severe Pain at 48 Hours After Surgery
Description: The proportion of patients reporting severe pain, defined as pain score (7-10) through the second postoperative day
Time Frame: 48 hours
Measure: Number; unit: percentage of patients with severe pain
Arm/Group | Single Shot Adductor Canal Block | 24 Hour Continuous Adductor Canal Block | 48 Hour Continuous Adductor Canal Block
Number analyzed (Participants) | 53 | 51 | 52
percentage of patients with severe pain | 21 | 14 | 12

2. Secondary Outcome: Pain Scores at 48 Hours After Surgery
Description: Average pain scores 48 hours after surgery. The scale used is the numeric rating pain scale. The scale values range from 0-10/ where 0 is no pain and 10 is the worst pain possible imagined on this scale
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale ( Pain score)
Arm/Group | Single Shot Adductor Canal Block | 24 Hour Continuous Adductor Canal Block | 48 Hour Continuous Adductor Canal Block
Number analyzed (Participants) | 53 | 51 | 52
units on a scale ( Pain score) | 5 (2) | 4.3 (2.5) | 3.9 (2.4)

3. Secondary Outcome: Functional Recovery After Surgery
Description: Cumulative ambulation distance in the second postoperative day measured in feet
Time Frame: 48 hours
Population: cumulative ambulation distance in second day after surgery
Measure: Median (Inter-Quartile Range); unit: Feet
Arm/Group | Single Shot Adductor Canal Block | 24 Hour Continuous Adductor Canal Block | 48 Hour Continuous Adductor Canal Block
Number analyzed (Participants) | 53 | 51 | 52
Feet | 155 [62 to 240] | 150 [70 to 240] | 200 [90 to 270]

4. Secondary Outcome: Patient-oriented Outcomes
Description: Quality of recovery (QoR)-9 score on the second day after surgery. This score is a result of a 9 item questionnaire. Answers to each item/question is scored as (0-1-2). The wort score a patient get in the questionnaire is 0 and the best score is 18, depending on the answer of each of the 9 questions and the sum of the scores of these answers
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale ( QoR score)
Arm/Group | Single Shot Adductor Canal Block | 24 Hour Continuous Adductor Canal Block | 48 Hour Continuous Adductor Canal Block
Number analyzed (Participants) | 53 | 51 | 52
units on a scale ( QoR score) | 12 [11 to 14] | 13 [11 to 15] | 13 [12 to 15]

ADVERSE EVENTS:
Arm/Group | Single Shot Adductor Canal Block | 24 Hour Continuous Adductor Canal Block | 48 Hour Continuous Adductor Canal Block
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes